CLINICAL TRIAL: NCT04911127
Title: Randomized, Double Blind, Placebo-Controlled Trial to Evaluate the Safety and Tolerability of Cannabidiol (CBD) in Moderate to Severe Rheumatoid Arthritis
Brief Title: Therapeutic Response of Cannabidiol in Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Veena Ranganath, MD, MS, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 19-01551; P64-01-003 (Other Grant/Funding Number: CMCR)
Record Dates: First submitted 2021-05-14; First posted 2021-06-02 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Rheumatoid Arthritis; Cannabis
MeSH Terms: conditions — Arthritis, Rheumatoid; Marijuana Abuse

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Participants will take capsules containing medium chain triglyceride (MCT) oil
  Interventions: Drug: Placebo capsules
- 200mg CBD twice daily (Experimental): Participants will take capsules containing cannabidiol amounting to 200mg CBD twice daily
  Interventions: Drug: 200mg Cannabidiol by capsules twice daily
- 400 mg CBD twice daily (Experimental): Participants will take capsules containing cannabidiol amounting to 400mg CBD twice daily
  Interventions: Drug: 400mg Cannabidiol by capsules twice daily

INTERVENTIONS:
Drug: 200mg Cannabidiol by capsules twice daily — 200mg twice daily via 50mg capsules
  Other Names: CBD
  Arms: 200mg CBD twice daily
Drug: 400mg Cannabidiol by capsules twice daily — 400mg twice daily via 50mg capsules
  Other Names: CBD
  Arms: 400 mg CBD twice daily
Drug: Placebo capsules — MCT oil capsules as placebo for CBD
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
The study will randomly assign Rheumatoid Arthritis (RA) patients on stable RA therapy to either placebo or cannabidiol (CBD). The overall goal of this proposal is to examine the efficacy and safety of CBD treatment as adjunctive to the medical management of RA patients.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double-blind clinical trial at the University of California, Los Angeles evaluating the efficacy, safety, and tolerability of oral cannabidiol (CBD) as adjunctive for rheumatoid arthritis (RA) patients on stable therapy. Patients with moderate to severe RA meeting study inclusion criteria will be randomly assigned to one of three treatment groups (CBD 200 mg BID, CBD 400 mg BID, or placebo). Patients in all groups will receive CBD or placebo under observation for 12 weeks with an additional follow-up phone call occurring 4 weeks after.

ELIGIBILITY:
Inclusion Criteria:

* Meet the American College of Rheumatology/European League Against Rheumatism (ACR/EULAR) 2010 Classification Criteria for Rheumatoid Arthritis
* Disease activity score (DAS28) >= 3.2
* Age >= 18
* Stable RA therapy for 12 weeks prior to baseline
* Power Doppler Score >= 5 (for the PDUS 34 joint score)
* Must use at least one highly effective method of contraception
* Written informed consent

Exclusion Criteria:

* Prior exposure to cannabis <= 28 days prior to baseline
* Current diagnosed substance use disorders (including Alcohol Use Disorder)
* Moderate (Child-Pugh B) or severe (Child-Pugh C) hepatic impairment
* Chronic infections
* >10mg of prednisone daily use
* Daily use of central nervous system (CNS) depressant medications (e.g. sedatives, hypnotics [zolpidem, temazepam, alprazolam, lorazepam, diphenhydramine etc.])
* Women who are pregnant, planning to become pregnant, or breast feeding
* Sexually active subjects and their partners who are of childbearing potential (ie, neither surgically sterile nor postmenopausal) and not agreeing to use adequate contraception
* Deemed unsafe by the investigator
* History of an allergic reaction or adverse reaction to cannabis is exclusionary.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2021-10-05 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Disease Activity Score (DAS28/ESR) | Baseline, 12 Weeks
  The DAS28 is a combined index for measuring disease activity in rheumatoid arthritis (RA). The index includes swollen joint counts (SJC) and tender joint counts (TJC), both scored 0-28 (higher scores indicate higher disease activity), as well as acute phase response (APR) determined as erythrocyte sedimentation rate (ESR), and general health (GH), both scored 1-100 (higher scores indicate higher disease activity). DAS28 was calculated according to the following formula: DAS28 equals (=) [0.56 multiplied by (*) the square root (√) of TJC] plus (+) [0.28 * √ of SJC] + (0.70 * the natural logarithm (ln) ESR in millimeters per hour (mm/h)] + [0.014 * GH in mm visual analogue assessment (VAS)]. A negative change from randomization indicated improvement.
Tolerability as assessed by participant attrition | 12 weeks
  Tolerability will be evaluated based on the number of participants that drop out due to treatment emergent adverse events or serious adverse events.

SECONDARY OUTCOMES:
Change in Power Doppler Synovitis Score (PDUS) | Baseline, 12 weeks
  34 joints will be evaluated using a 0 to 3 point scale for each joint and the sum of these represents PDUS. PDUS ranges from 0 to 102. Scores of 0 indicate the least amount of inflammation of the joint while scores of 3 indicate the most amount of inflammation. A higher value of the total score for PDUS represents more severe disease level.
Change in Grey Scale Synovial Hypertrophy Score (GSUS) | Baseline, 12 weeks
  34 joints will be evaluated using a 0 to 3 point scale for each joint and the sum of these represents GSUS. GSUS ranges from 0 to 102. Scores of 0 indicate the least amount of inflammation of the joint while scores of 3 indicate the most amount of inflammation. A higher value of the total score for GSUS represents more severe disease level.

OTHER OUTCOMES:
Change in inflammatory cytokine and chemokine concentrations | Baseline, 12 weeks
  Inflammatory cytokines and chemokine concentrations from plasma will be evaluated using multiplex cytokine array.
Change in white blood cell (WBC) subset percentages | Baseline, 12 weeks
  WBC subset percentages will be assessed via flow cytometry.
Change in Clinical Disease Activity Index (CDAI) | Baseline, 12 weeks
  CDAI was derived as the sum of the following: tender joint count (TJC), swollen joint count (SJC), participant global assessment (PGA) of disease activity, and physician assessment of disease activity. TJC and SJC were taken as the number of tender and swollen joints, respectively, out of 28 assessed joints. PGA and physician assessment of disease activity were scored 0-100 millimeters (mm) and rounded to the nearest centimeter (cm) on a visual analog scale (VAS), where higher scores indicate greater perceived disease activity. The total CDAI score range is 0-76, where higher scores indicate increased disease activity.
Change in Health Assessment Questionnaire - Disability Index (HAQ-DI) | Baseline, 12 weeks
  The HAQ-DI is a patient-reported assessment of physical function that includes 20 items in eight categories representing a comprehensive set of functional activities, including dressing and grooming, arising, eating, walking, hygiene, reach, grip and common daily activities. Patients are asked about their ability to complete these tasks in the past week using the following categories: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). Scores on each task are summed and averaged to provide an overall score ranging from 0 (best) to 3 (worst), with a higher score representing a high-dependency disability.

CONTACTS AND LOCATIONS:
Overall Officials: Ziva Cooper, PhD, Principal Investigator — University of California, Los Angeles; Veena Ranganath, MD, MS, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA David Geffen School of Medicine, Division of Rheumatology, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No